CLINICAL TRIAL: NCT03271619
Title: Electrical Safety of Rescuers in Contact With Patients During Implanted Cardioverter Defibrillator Discharge
Brief Title: Electrical Safety of Implantable Cardioverter Defibrillators
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13/SC/0427
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Defibrillators, Implantable; Cardiac Arrest
Keywords: Safety Issues
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transvenous ICD: Patients with a transvenous ICD undergoing defibrillation testing.
  Interventions: Other: Surface current measurement
- Subcutaneous ICD: Patients with a subcutaneous ICD undergoing defibrillation testing.
  Interventions: Other: Surface current measurement

INTERVENTIONS:
Other: Surface current measurement — Measurement of surface current between electrodes placed on the chest wall during defibrillation

SUMMARY:
Patients at risk of developing life-threatening heart rhythms may require the implantation of a small device called a cardioverter-defibrillator (ICD), which constantly monitors the heart rhythm and delivers an electrical shock to the heart when indicated, in order to return the heart back to a normal rhythm. Many thousands of these devices have been implanted and are electrically active in patients who collapse and need resuscitation.

When a patient with an ICD collapses, the device may discharge without warning while a rescuer is performing external chest compressions (cardiac massage). Conventional ICDs placed below the left collar bone typically deliver 35-50 J energy when they discharge, but newer ICDs placed under the skin (S-ICD) alongside the breastbone deliver a larger energy when discharging; typically 50-80J energy.

Rescuers performing external chest compressions on a patient during conventional ICD discharge have reported the sensation of a painful electrical shock and permanent nerve damage. In these situations, rescuers appear to have been exposed to electrical current from the ICD considerably in excess of that which is considered a safe threshold.

Studies of surface current resulting from discharge of conventional ICDs have been reported in excess of 100 mA which is far in excess of the safe 1 mA limit, and puts the rescuer at considerable risk of tissue damage and possible dangerous heart rhythms. The newer S-ICDs deliver approximately 50% more energy and have the potential to result in exposure of a rescuer to even higher currents.

With increasing numbers of the S-ICDs being implanted, and the inevitability that rescuers will soon find themselves exposed to leakage current from these devices, there is a need to examine the leakage currents arising from these devices and assess any subsequent risk to a rescuer performing external chest compressions.

DETAILED DESCRIPTION:
Rationale for Study:

When patients undergo elective implantation of an ICD, the device is tested by inducing ventricular fibrillation (VF) in the patient and allowing the ICD to sense, charge and discharge in an attempt to shock the patient back into a normal rhythm. This provides a controlled, elective situation in which to measure the cutaneous current on the patient's skin which is the current to which a rescuer could potentially be exposed.

By understanding the leakage currents from these devices, the investigators will be able to better understand the safety of rescuers in contact with patients fitted with an ICD and make specific recommendations to enable to safe undertaking of uninterrupted external chest compressions while the ICD may be discharging.

STUDY OBJECTIVES

Primary Objective:

To measure cutaneous leakage current on the chest wall during conventional and S-ICD discharge.

Secondary Objectives:

To make recommendations based on this data regarding the safety of rescuers in contact with a patient during ICD discharge.

ENDPOINTS

Primary Endpoint:

Maximum cutaneous current measured at multiple sites on the chest wall during ICD discharge.

STUDY DESIGN This is a prospective cohort study, aiming to study sequential patients undergoing elective ICD implantation and testing over a 12 month period at University Hospital Southampton.

The patient will undergo elective ICD implantation according to normal protocol. There will be no change in their treatment. After induction of general anaesthesia, an array of small self-adhesive electrodes (similar to ECG 'dots') will be placed on the patient's chest wall, and connected to a multichannel recording device.

After implantation of the ICD, the device will be tested as per normal protocol. VF is induced in the patient. The ICD senses this arrhythmia, charges and immediately delivers a shock to the myocardium. As this shock is delivered, the investigators will record the current reaching the surface electrode array using the multichannel recorder. Most patients only require one shock as defibrillation rates with ICDs are >90%. If a second shock is required, the ICD will charge automatically and discharge once again. If this occurs, the investigators will also measure the cutaneous current at this second, higher energy level. The study is then concluded. Any subsequent shocks are delivered through external paddles and the investigators would not require any data from this stage of the procedure.

STUDY POPULATION Number of Participants The investigators aim to assess 20 patients undergoing conventional ICD implantation and a further 20 patients undergoing S-ICD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with implanted defibrillators (ICDs) undergoing defibrillation testing
* Patients undergoing ICD implantation that requires a defibrillation test at the end of the implantation.

Exclusion Criteria:

* Enrolment in other ICD-related studies
* Patients <18 yrs age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with implanted defibrillators (ICDs) undergoing defibrillation testing.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Surface current during defibrillation | Approximately 10 mSec as the ICD discharges (i.e. at the time of testing)
  To measure cutaneous leakage current on the chest wall during conventional and S-ICD discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Deakin, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Please contact researchers directly

REFERENCES:
- [Background] Willcox ME, Prutkin JM, Bardy GH. Recent developments in the subcutaneous ICD. Trends Cardiovasc Med. 2016 Aug;26(6):526-35. doi: 10.1016/j.tcm.2016.03.004. Epub 2016 Mar 15. PMID 27079889
- [Background] Chue CD, Kwok CS, Wong CW, Patwala A, Barker D, Zaidi A, Mamas MA, Cunnington C, Ahmed FZ. Efficacy and safety of the subcutaneous implantable cardioverter defibrillator: a systematic review. Heart. 2017 Sep;103(17):1315-1322. doi: 10.1136/heartjnl-2016-310852. Epub 2017 Jul 7. PMID 28687562
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Clements PA. Hazards of performing chest compressions in collapsed patients with internal cardioverter defibrillators. Emerg Med J. 2003 Jul;20(4):379-80. doi: 10.1136/emj.20.4.379. No abstract available. PMID 12835365
- [Background] Stockwell B, Bellis G, Morton G, Chung K, Merton WL, Andrews N, Smith GB. Electrical injury during "hands on" defibrillation-A potential risk of internal cardioverter defibrillators? Resuscitation. 2009 Jul;80(7):832-4. doi: 10.1016/j.resuscitation.2009.04.010. Epub 2009 May 14. PMID 19446388
- [Background] Niwano S, Kojima J, Inuo K, Saito J, Kashiwa T, Suyama M, Toyoshima T, Aizawa Y, Izumi T. Measurement of body surface energy leakage of defibrillation shock by an implantable cardioverter defibrillator. Pacing Clin Electrophysiol. 2002 Aug;25(8):1212-8. doi: 10.1046/j.1460-9592.2002.01212.x. PMID 12358172